CLINICAL TRIAL: NCT02063841
Title: A Prospective Double-blind, Randomized, Sham-controlled Trial to Evaluate the Effect of a Lead Free Drape on Scatter Radiation Exposure to Endoscopy Staff During Endoscopic Retrograde Cholangiopancreatography
Brief Title: Digestive Endoscopy Suite Radiation Controlling Protective Strategies
Acronym: D-ERCP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1210010994.Jamidar
Record Dates: First submitted 2014-02-12; First posted 2014-02-14 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Radiation Exposure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sterile identical sham drape (Active Comparator): Sham drape and conventional protection (wearing a lead apron and thyroid shield as well as suspension of a standard lead skirt over the X-ray source).
  Interventions: Device: sterile identical sham drape
- lead-free protective drape containing bismuth and antimony (Experimental): lead-free protective drape containing bismuth and antimony (RADPAD®) hung around the fluoroscopy image intensifier to prevent scatter radiation, and conventional protection (wearing a lead apron and thyroid shield as well as suspension of a standard lead skirt over the X-ray source).
  Interventions: Device: lead-free protective drape containing bismuth and antimony (RADPAD®)

INTERVENTIONS:
Device: lead-free protective drape containing bismuth and antimony (RADPAD®)
  Arms: lead-free protective drape containing bismuth and antimony
Device: sterile identical sham drape
  Arms: sterile identical sham drape

SUMMARY:
ERCP is associated with radiation exposure to the endoscopist and staff, which may be significant at high volume programs despite the use of lead aprons. We hypothesize that draping of the fluoroscopy image intensifier may significantly reduce staff radiation exposure and help achieve implementation of the ALARA (As Low As Reasonably Achievable) principle.

DETAILED DESCRIPTION:
A total of 100 consecutive ERCP procedures were randomly assigned to the radiation-attenuating or sham drape in a 1:1 ratio. There were 2 subjects, the endoscopists performing ERCP and the nurse assisting in the procedure.

ELIGIBILITY:
Inclusion Criteria:

* All the ERCP procedures done by the same endoscopist and nurse are enrolled
* Patients age >19

Exclusion Criteria:

* Fluoroscopic procedures other than ERCP were excluded.

Ages: 45 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Amount of radiation exposure | Length of Endoscopic retrograde cholangiopancreatography, average 5 minutes
  Comparing the use of a lead-free protective drape containing bismuth and antimony and a sterile sham protective drape, radiation dose (RD) was measured at 3 different sites (endoscopist's eye (1) and thyroid (2), and assisting nurse's thyroid (3)) with personal dosimeters placed outside of eyeglass frames and the thyroid shield. The unit of measurement is each event. The subject was subjected to radiation during 100 Endoscopic retrograde cholangiopancreatography procedures.Both groups used standard of care lead protection.

SECONDARY OUTCOMES:
Estimate cumulative annual radiation risk | Length of Endoscopic retrograde cholangiopancreatography, average 5 minutes
  Comparing the use of a lead-free protective drape containing bismuth and antimony and a sterile sham protective drape, radiation dose (RD) was measured at 3 different sites (endoscopist's eye (1) and thyroid (2), and assisting nurse's thyroid (3)) with personal dosimeters placed outside of eyeglass frames and the thyroid shield. The unit of measurement is each event. The subject was subjected to radiation during 100 endoscopic retrograde cholangiopancreatography procedures. The cumulative estimated annual absorbed radiation dose was estimated from the data collected during the study time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Jamidar, MD, Principal Investigator — Yale University
Locations (1):
- Endoscopy Center, Smilow Cancer Center, Yale New Haven Hospital, New Have, Connecticut, United States

REFERENCES:
- See also: A Double-Blind, Randomized, Sham-Controlled Trial of the Effect of a Radiation-Attenuating Drape on Radiation Exposure to Endoscopy Staff During ERCP — http://www.nature.com/ajg/journal/vaop/ncurrent/full/ajg201585a.html